CLINICAL TRIAL: NCT02726945
Title: Use of Autologous Adipose-Derived Stromal Vascular Fraction to Treat Osteoarthritis of the Knee: A Controlled, Randomized, Double-Blinded Trial
Brief Title: Adipose-derived SVF for the Treatment of Knee OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GID BIO, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GIDOA-01
Record Dates: First submitted 2016-03-24; First posted 2016-04-04 (Estimated); Results first posted 2019-08-21 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2020-02

CONDITIONS: Osteoarthritis (OA)
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low Dose SVF (Experimental): This group of subjects will receive a low dose of SVF for treatment of knee OA.
  Interventions: Device: GID SVF-2
- High Dose (Experimental): This group of subjects will receive a high dose of SVF for treatment of knee OA.
  Interventions: Device: GID SVF-2
- Placebo (Placebo Comparator): This group of subjects will receive a placebo with no SVF Cells for treatment of knee OA.
  Interventions: Other: Placebo

INTERVENTIONS:
Device: GID SVF-2 — The GID SVF-2 device is a sterile single-use disposable canister used for harvesting, filtering, separating, and concentrating autologous stromal vascular fraction cells from adipose tissue for reintroduction to the same patient during a single surgical procedure for treatment of pain associated with joint osteoarthritis.
  Arms: High Dose; Low Dose SVF
Other: Placebo — Placebo Control
  Arms: Placebo

SUMMARY:
This is a pivotal study. The study will examine the safety and efficacy of autologous adipose-derived stromal vascular fraction (SVF) cells processed with the GID SVF-2 device for pain, function and stiffness in the knees of osteoarthritic subjects.

DETAILED DESCRIPTION:
Osteoarthritis is the main form of arthritis and affects over 20 million people in the United States. In the knee it can cause severe pain, reduced functionality and increased stiffness thus, a treatment that would reduce pain, increase function and reduce stiffness would be of benefit to many people.

This study will collect and disassociate adipose tissue and inject the stromal vascular fraction into the knee of the same patient. The study is controlled, randomized and double-blinded with 2 SVF treatments (high and low dose) and a placebo control.

ELIGIBILITY:
Inclusion Criteria:

* Grade II or Grade III osteoarthritis using Kellgren-Lawrence grading scale (K-L Grade) as diagnosed using weight bearing X-ray, physician review, and/or pre-op MRI.
* Study Subjects must have failed a minimum of at least two conservative therapies, spanning a period of at least 3 months.
* Study Subjects must be willing to voluntarily give written Informed Consent to participate in the study and sign the Health Insurance Portability and Accountability Act (HIPAA) authorization before any study procedures are performed.
* Subjects will be in good health (ASA Class I-II) with a BMI < 35.
* Subjects must have continued pain in the knee despite conservative therapies for at least 3 months.
* Subjects with unilateral disease must present with symptomatic knee pain using the WOMAC subscale for pain.
* Subjects must speak, read and understand English.
* Subjects must be reasonably able to return for multiple follow-up visits.

Exclusion Criteria:

* Subjects whose knee pain is caused by, (i) diffuse edema, (ii) displaced meniscus tear, (iii) lesion greater than 1 cm in any direction, or (iv) osteochondritis dissecans.
* Subjects who have had surgery of either knee within 6 months prior to the screening visit.
* Subjects who have had a major injury to the targeted knee within 12 months prior to enrolling in the study.
* Subjects who have had an injection in either knee in the prior 3 months, including corticosteroids, viscosupplementation or platelet rich plasma (PRP).
* Subjects who have gout, rheumatoid arthritis, lupus arthropathy, psoriatic arthritis, avascular necrosis, severe bone deformity, infection of the knee joint, fibromyalgia, pes anserine bursitis, or neurogenic or vascular claudication.
* Subjects who have symptomatic OA of the hips, spine, or ankle that would interfere with the evaluation of the treated knee.
* Subjects that are unwilling to stop taking prescription or over the counter pain medication for 7 days prior to any visit
* Subjects that are allergic to lidocaine, epinephrine or valium
* Subjects with a history of bleeding disorders, anticoagulation therapy that cannot be stopped as prior to injection.
* Subjects with systemic immunosuppressant use within six (6) weeks from screening and subjects with HIV/viral hepatitis.
* Subjects with chondrocalcinosis, Paget's disease and Villonodular synovitis
* Subjects that use any form of tobacco
* Women that are pregnant or planning to become pregnant during the study.
* Subjects on long term use of oral steroids
* History of any chemotherapy or radiation therapy of the targeted/treatment leg or adipose harvest site.
* Subjects currently on worker's compensation

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2019-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Good, PhD, Study Director — GID BIO, Inc.
Locations (3):
- United States (3):
  - Cooper University Hospital, Camden, New Jersey
  - Rothman Institute, Egg Harbor, New Jersey
  - Texas Plastic Surgery, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
This study will report average demographics and WOMAC OA score. Individual adverse events may be reported.

REFERENCES:
- [Background] Fodor PB, Paulseth SG. Adipose Derived Stromal Cell (ADSC) Injections for Pain Management of Osteoarthritis in the Human Knee Joint. Aesthet Surg J. 2016 Feb;36(2):229-36. doi: 10.1093/asj/sjv135. Epub 2015 Aug 3. PMID 26238455
- [Background] Garza GR, Palomera T, Dumanian GA and Dos-Anjos S. Use of Autologous Adipose-derived Stromal Vascular Fraction to Treat Osteoarthritis of the Knee: A Feasibility and Safety study. J Regen Med. 2015;4(1)
- [Derived] Garza JR, Campbell RE, Tjoumakaris FP, Freedman KB, Miller LS, Santa Maria D, Tucker BS. Clinical Efficacy of Intra-articular Mesenchymal Stromal Cells for the Treatment of Knee Osteoarthritis: A Double-Blinded Prospective Randomized Controlled Clinical Trial. Am J Sports Med. 2020 Mar;48(3):588-598. doi: 10.1177/0363546519899923. PMID 32109160

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment opened April 2015 and the first subject was enrolled in the study in July 2016. Recruitment was completed in September 2017.
Groups:
- Low Dose SVF: This group of subjects will receive a low dose of SVF (15 ± 2.5 x 10e6 SVF cells) for treatment of knee OA.
- High Dose SVF: This group of subjects will receive a high dose of SVF (30 ± 2.5 x 10e6) SVF cells for treatment of knee OA.
- Placebo: This group of subjects will receive a placebo with no SVF (0 SVF cells) for treatment of knee OA.
Period: Overall Study
Arm/Group | Low Dose SVF | High Dose SVF | Placebo
Started | 13 | 13 | 13
Completed | 13 | 12 | 12
Not Completed | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Elected to have total knee replacement | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose SVF | High Dose SVF | Placebo | Total
Number analyzed (Participants) | 13 | 13 | 13 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (7.9) | 59.5 (11.7) | 57.1 (9.1) | 59.0 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 7 | 22
  Male | 4 | 7 | 6 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3 | 6
  Not Hispanic or Latino | 12 | 11 | 10 | 33
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 13 | 13 | 12 | 38
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 13 | 39
Kellgren Lawrence Osteoarthritis Grade [Count of Participants; unit: Participants] — Kellgren-Lawrence Osteoarthritis Scale
  * Grade 0, None - No radiographic features of OA are present
  * Grade 1, Doubtful - Doubtful narrowing of joint space and possible osteophytic lipping
  * Grade 2, Minimal - Definite osteophytes and possible narrowing of joint space on anteroposterior weight-bearing radiograph
  * Grade 3, Moderate - Moderate multiple osteophytes, definite narrowing of joint space and some sclerosis and possible deformity of bone ends
  * Grade 4, Severe - Large osteophytes, marked narrowing of joint space, severe sclerosis and definite deformity of bone ends
  Participants
    KL Grade II | 4 | 4 | 4 | 12
    KL Grade III | 9 | 9 | 9 | 27

OUTCOME MEASURES:

1. Primary Outcome: Safety - Number of Participants With Treatment-Emergent Serious Adverse Events
Description: Subjects will be monitored for serious and device related adverse events. Baseline MRIs will be compared to 1 year for any abnormal findings.
Time Frame: up to 1 year
Population: Thirty-eight subjects were monitored to 1 year. One subject was monitored for 6 weeks, when the subject withdrew from the study to receive a total knee replacement.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose SVF | High Dose SVF | Placebo
Number analyzed (Participants) | 13 | 13 | 13
Participants
  Serious Adverse Events | 0 | 0 | 0
  Device Related Serious Adverse Events | 0 | 0 | 0
  MRI abnormalities | 0 | 0 | 0

2. Secondary Outcome: Efficacy - Percent Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Score From Baseline to 6 Months
Description: The primary efficacy will be achieved if either dose group is shown to be superior to the placebo group at 6 months post-treatment, using the percent change in WOMAC score from baseline as the primary variable.
  The WOMAC score consists of 3 subscales, pain, stiffness and function. The overall score is normalized to a range of 0 to 100 points with a lower score indicating less symptoms of osteoarthritis.
Time Frame: baseline and 6 months
Population: The data set was analyzed with an Intent-to-treat principle and used the last observation carried forward (LOCF) method for missing data.
Measure: Median (Inter-Quartile Range); unit: percentage of change in WOMAC score
Arm/Group | Low Dose SVF | High Dose SVF | Placebo
Number analyzed (Participants) | 13 | 13 | 13
percentage of change in WOMAC score | 52 [29 to 88] | 84 [19 to 91] | 25 [-25 to 58]
Statistical Analysis 1: Comparison: Low Dose SVF vs Placebo; Data from the groups showed a strong non-normal distribution, thus non-parametric methods were used with a Bonferroni correction for multiple comparison . Statistical significance was defined as either of the treatment groups to be superior to the placebo group; Test type: Superiority; p = 0.023, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: High Dose SVF vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.043, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Low Dose SVF | High Dose SVF | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 1/13 | 2/13 | 0/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose SVF (N=13) | High Dose SVF (N=13) | Placebo (N=13)
Swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Swelling of the knee that resolved spontaneously
Possible Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) — Sterility test showed 1 suspicious colony at 3 days. The patients showed no sign of infection.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT02726945/Prot_SAP_000.pdf